CLINICAL TRIAL: NCT01914627
Title: A Single-centre Randomised, Active-controlled, Observer-blinded, Parallel Group Trial to Evaluate the Efficacy and Safety of a Topical Dimeticone Formulation (Loion®) Compared to 10% Salicylic Acid in the Removal of Scaling in Patients With Chronic Psoriasis Capitis
Brief Title: Parallel Group Trial to Evaluate the Efficacy and Safety of Loion® Compared to 10% Salicylic Acid in Patients With Chronic Psoriasis Capitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G. Pohl-Boskamp GmbH & Co. KG (Industry)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0741/179
Record Dates: First submitted 2013-07-17; First posted 2013-08-02 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-02

CONDITIONS: Scalp Psoriasis
Keywords: Psoriasis capitis; Scaling; Salicylic acid; Dimethicone; Plaque removal
MeSH Terms: interventions — dimethicone; Salicylic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loion (Experimental)
  Interventions: Drug: Dimethicone
- SA-Gel (Active Comparator)
  Interventions: Drug: Salicylic Acid

INTERVENTIONS:
Drug: Dimethicone — The treatment will be carried out once daily (in the evening) onto all scaling areas of the scalp over a period of 2 weeks, with the last application of investigational products being applied one day prior to the final visit.
  Arms: Loion
Drug: Salicylic Acid — The treatment will be carried out once daily (in the evening) onto all scaling areas of the scalp over a period of 2 weeks, with the last application of investigational products being applied one day prior to the final visit.
  Arms: SA-Gel

SUMMARY:
The study will be conducted to evaluate the efficacy and safety of a topical dimeticone formulation (Loion®) compared to 10% salicylic acid in octyl-dodecanol with 15% Macrogol-4-laurylether for the removal of scaling in patients with chronic psoriasis capitis (scalp psoriasis).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Having a diagnosis of chronic psoriasis capitis (scalp psoriasis) with or without the involvement of other body areas and with or without psoriatic arthritis.
* PSSI ≥5 (range 0-72)
* Scaling ≥2 (on an scale from 0 to 4)
* At least 10% of scalp area affected
* If a women:
* Postmenopausal
* Premenopausal and using an established oral, injected or implanted hormonal method of contraception, intrauterine device (IUD) or intrauterine system (IUS)
* Negative pregnancy test at inclusion
* Patients with no concomitant systemic psoriasis medication.
* Willingness and adherence to the prohibitions and restrictions specified in the study protocol.
* Willingness to self-administer the drug.
* Signed informed consent document indicating that the patient to be included understands the purpose of and the procedures for the study and is willing to participate.

Exclusion Criteria:

* Patients having a solely non- plaque form of psoriasis (e.g. erythrodermic, guttate, pustular).
* Patients with uncontrolled psoriasis under the current treatment.
* Patients having received topical keratolytic agents for the scalp within the past 2 weeks and topical steroids for the scalp within the past week (prior to inclusion).
* Patients receiving systemic antipsoriatic drugs, immunosuppressants or systemic corticosteroids (within 4 weeks prior to inclusion).
* Women who are pregnant or breastfeeding or planning to become pregnant during the observational period.
* Patients participating in another study using an investigational agent or procedure during participation in the study observation period.
* Known hypersensitivity to any ingredient in the investigational products' formulations.
* Having any condition that in the opinion of the investigator makes the participation not be in the best interest of the subject.
* Employees and staff of the investigator or study site with direct involvement in the study as well as family members of the employee or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Scaling | at Day 7
  To evaluate improvement of scaling of patients exposed to Loion or standard therapy for psoriasis capitis

SECONDARY OUTCOMES:
Psoriasis Scalp Severity Index (PSSI) | at Day 0, day 3, day 7, day 14
  To evaluate clinical outcome of patients exposed to Loion or standard therapy for psoriasis capitis

OTHER OUTCOMES:
Psoriasis Area Severity Index (PASI) | at Day 0, day 3, day 7, day 14
  To evaluate clinical outcome of patients exposed to Loion or standard therapy for psoriasis capitis
Body Surface Area (BSA) | at Day 0, day 3, day 7, day 14
  To evaluate clinical outcome of patients exposed to Loion or standard therapy for psoriasis capitis
Physician Global Assessment (PGA) | at Day 0, day 3, day 7, day 14
  To evaluate global severity of skin of patients exposed to Loion or standard therapy for psoriasis capitis
Scalp Physician Global Assessment (sPGA) | at Day 0, day 3, day 7, day 14
  To evaluate global severity of scalp skin of patients exposed to Loion or standard therapy for psoriasis capitis
Dermatology Life Quality Index (DLQI) | at Day 0, day 3, day 7, day 14
  To evaluate disease related quality of life of patients exposed to Loion or standard therapy for psoriasis capitis
Patient Benefit Index (PBI) | at Day 0, day 3, day 7, day 14
  To evaluate the patient benefit of Loion or standard therapy for psoriasis capitis
EuroQol Questionnaire (EQ-5D) | at Day 0, day 3, day 7, day 14
  To evaluate general state of health of patients exposed to Loion or standard therapy for psoriasis capitis
Adverse and serious adverse events | 14 days
  Risk for adverse events and serious adverse events for patients exposed to Loion or standard therapy for psoriasis capitis

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Augustin, Prof., Principal Investigator — University Medical Center Hamburg-Eppendorf (UKE)
Locations (1):
- University Medical Center Hamburg-Eppendorf (UKE), Hamburg, Germany